| Official Title of the Study: | A Phase 1, Randomized, Double-Blind, Placebo-<br>Controlled Study to Assess the Safety, Tolerability,<br>Pharmacokinetics, and Immunogenicity of REGN17092,<br>an Anti-SARS-CoV-2 (COVID-19) Monoclonal Antibody,<br>in Adult Healthy Volunteers |
|---|---|
| EU CT: | 2023-505041-52-00 |
| Protocol Number: | R17092-HV-2312 |
| Sponsor of the Study: | Regeneron Pharmaceuticals, Inc. 777 Old Saw Mill River Road Tarrytown, NY 10591 United States |
| European Representative: | One Warrington Place Dublin 2, DO2 HH27 Ireland |
| Site Name: | Center for Clinical Pharmacology, UZ Leuven |
| Main Address of Site: | Campus Gasthuisberg, Herestraat 49, B-3000 Leuven, Belgium |
| Local Investigator (Study doctor): | dy Prof. Dr. Jan de Hoon |

# Who can I contact in case of questions?

| Name | Function In case of | | Contact details |
|---|---|---|---|
| De Hoon, Jan | Principal<br>Investigator of the<br>site | Information, problems, or concerns | 016 34 20 20<br>ckf@uzleuven.be |
| | The trial staff | Information, problems, or concerns | 016 34 20 20 |
| | Emergency contact | Emergency | 0479 88 08 71<br>0472 72 23 68 |
| | Patient rights<br>ombudsman | Concerns relating to your rights as a participant in a trial | Ombudsdienst<br>016 34 48 18 |
| Name and address of insurance company of the sponsor & contact of insurer | company of the sponsor disagreement or complaint on a damage claim tof | | Chubb European Group SE, Avenue Louise 480, 1050 Brussels, Belgium pc.operations.benelux@chubb.com chubb.com/benelux +31(0)102893545 Policy N°: BECANY02059 |
| confidentia | | Questions<br>relating to the<br>confidentiality<br>of your data | E-mail: privacy@kuleuven.be |
| | Belgian Data Protection Authority Complaints relating to the confidential of your data | | 32 2 274 48 00<br>E-mail: contact@apd-gba.be |

# CHAPTER I – DESCRIPTION OF THE STUDY AND YOUR RIGHTS WHEN PARTICIPATING

# 1. Why are we doing this study?

This study will evaluate the investigational medicinal product, REGN17092 (called "study drug" in this form). An investigational medicinal product is a medicinal product that is still being studied to evaluate its efficacy, safety, or mode of action.

The information obtained during this study may contribute to a better understanding of the use of the study drug or to the development of a new medicinal product for the treatment of coronavirus disease 2019 (COVID-19).

The purpose of this study is to learn about the safety and tolerability of different doses of REGN17092 administered with a needle either under the skin (subcutaneous) as an injection or into a vein (intravenous) as an infusion in healthy participants. This is the first time that REGN17092 will be given to people.

Other aims are to assess:

- how much of the study drug is in the blood at different times
- whether the body makes its own antibodies against the study drug (which could make the drug less effective or lead to side effects)

REGN17092 is a monoclonal antibody. Antibodies are made by your immune system to fight infections. A monoclonal antibody is made in a laboratory. Monoclonal antibodies can be developed to fight against specific infections, like infection from a virus.

COVID-19 is caused by a virus called severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). This virus uses a spike protein to attach to the cells it infects. The spike protein helps the virus infect cells in the nose, throat, lungs, and other tissues, leading to COVID-19 symptoms.

REGN17092 is designed to block the SARS-CoV-2 spike protein. When the spike protein is blocked, the virus may not be able to cause infection. This may prevent people from becoming infected. For those who are infected, this may prevent them from developing COVID-19 symptoms or stop symptoms from getting worse.

Viruses are always changing. There are now different variants (types) of the virus that causes COVID-19. Some of these variants may lead to worse disease, may be more contagious, or may be harder to treat or vaccinate against. REGN17092 was designed to work against variants, including Delta and Omicron.

REGN17092 is not authorized or approved by any government agency to treat or prevent COVID-19 or any other disease or condition.

The drug is considered investigational for the purposes described in this study.

Regeneron, its collaborators or those developing the trial drugs, and their affiliates, representatives, agents, and contractors (the "Regeneron Parties"), are involved in the study and may use the data and samples collected in the study to conduct the research described in this consent form.

R17092-HV-2312 Main ICF Version 2.0

# 2. Why am I being asked to take part?

This study is trying to understand the safety of REGN17092 in volunteers who are generally healthy and who have been vaccinated for COVID-19. You are being asked to participate in this study because you have been fully vaccinated against COVID-19. In order to join, you will also have to test negative for the virus that causes COVID-19. The study doctor or staff will discuss other requirements you will need to meet in order to enter the study.

# 3. Do I have to take part in a study?

Your participation in a study is voluntary and must remain free of any coercion. This means that you have the right not to take part in the study or to withdraw at any time without giving a reason, even if you previously agreed to take part. Your decision will not affect your relationship with the study doctor or your treating physician, nor will it affect the quality of your future medical care.

# 4. What will happen during the study?

This study will include up to 128 participants in Belgium.

This study is a randomized, double-blind, placebo-controlled study:

- "Double-blind" means that neither you nor the study doctor will know which treatment group you have been placed in (ie, if you are receiving the study drug [REGN17092] or placebo). This is done to make sure the results of the study cannot be influenced by anyone. If there is an urgent need, the study doctor can find out quickly which study medicine you are receiving.
- A "placebo" is an inactive substance that looks like the study drug REGN17092, but which contains no medicine. If you agree to take part in this study, you will receive either the study drug or placebo.
- "Randomized" means that the group you will be placed in is decided by chance, similar to drawing numbers out of a hat or flipping a coin. You will have a 3 in 4 (75%) chance of receiving REGN17092 and a 1 in 4 (25%) chance of receiving placebo.

# **Course of the Study**

The study consists of 3 periods:

- a screening period
- a treatment period
- a follow-up period with an end of study visit

Overall, your participation in the study will last about 365 days (excluding the screening period of up to 28 days) and involve up to 11 visits. At the discretion of the study doctor, additional visits may be required to monitor your health.

During each of the visits, several examinations or procedures will be required in connection with the study. These examinations or procedures are listed in CHAPTER III- STUDY CALENDARS at the end of this form.

# **Screening Period**

In the screening period, which is up to 28 days before administration of the study drug or placebo, you will be asked to come to the clinical study unit for initial screening to ensure that you are in good health and to see if you qualify for the study. This first visit is known as the screening visit (visit 1). During this visit, you will undergo several examinations.

Firstly, the study doctor or a member of the study staff will discuss the study and the requirements for participation in this study with you. It is important that you are completely truthful with the study doctor and study staff about your health history. You cannot participate in this study if you do not meet all requirements.

At the discretion of the study doctor, the screening procedures may be performed on different days during the screening period. This may increase the total number of clinical study unit visits. The study staff will discuss this with you.

When the results of the screening examinations are available, the study doctor, in accordance with the inclusion and exclusion criteria defined in the study protocol, will decide whether you can participate in the study and when you should return to the clinical study unit for the next study procedures.

You must inform the study staff immediately about any side effect or other discomforts you might experience during the whole study course, from the screening visit onwards.

#### **Treatment Period**

If you meet all the conditions required to be enrolled in the study according to the results from the screening period and agree to take part in the study, you will begin the treatment period and undergo further tests and examinations described in this form. If you have any side effects, the study doctor might determine that it is necessary to perform additional tests, which will be considered as specific to the study.

The study has up to 7 main study cohorts (groups) and may have up to 3 expansion cohorts for additional safety evaluation of the REGN17092 at 1 or more dose levels.

If you are assigned to one of the main study cohorts, you will be admitted to the clinical study unit the day before dosing or on the day of dosing, at the discretion of the study doctor. The study doctor or member of the study staff will discuss the procedures and samples needed when you get admitted to the clinical study unit. The results of these tests will determine whether you are still eligible to participate in the study.

You may be enrolled into one of 7 main study cohorts or one of the expansion cohorts. On day 1 of the treatment period, a single dose of the study drug (REGN17092) or placebo will be administered either under the skin or via an infusion in a vein. The study doctor will let you know if you are receiving the treatment under the skin or as an infusion in a vein before it is administered.

You will have a 3 in 4 (75%) chance of receiving REGN17092 and 1 in 4 (25%) chance of receiving placebo.

The <u>main study cohort</u> planned dose levels and route of administration are summarized in the table below. The planned doses may be decreased based on ongoing testing and/or safety and tolerability.

| Cohorts with treatment administered as an infusion in a vein | Dose of REGN17092 |
|---|---|
| 1 | 300 mg or placebo |
| 3 | 1200 mg or placebo |
| 5 | 2400 mg or placebo |
| 6 | Up to 150 mg or placebo |
| Cohorts with treatment administered under the skin | Dose of REGN17092 |
| 2 | 300 mg or placebo |
| 4 | 1200 mg or placebo |
| 7 | Up to 150 mg or placebo |

If you are in the main study cohort, you may be admitted to the clinical study unit the night before dosing (at the discretion of the study doctor) and will remain in the clinical study unit for at least 24 hours after dosing on day 1. On day 2, the study doctor will assess if you meet the discharge criteria based on a physical examination, vital signs, and monitoring of side effects. If you meet the discharge criteria, you may leave the clinical study unit and move to the follow-up period. If you do not meet the discharge criteria, you may be asked to remain at the clinical study unit for additional monitoring or to come back to the clinical study unit for additional visits. The study staff will discuss these criteria with you.

#### Dose Escalation

Doses of REGN17092 will be increased as summarized in the table above. The study doctor and sponsor will evaluate the safety and tolerability data. Once the administered dose level is considered to be safe by the sponsor and the study doctor, approval will be given for administration of the next dose level in the next cohort. If the study doctor and sponsor agree, adjustments of initially planned dose levels may be introduced without exceeding the highest dose indicated in the table above. If this occurs, the study doctor and/or study staff will discuss this with you. You will be informed if this happens.

# Sentinel Dosing

With the exception of cohorts 6 and 7, in order to monitor safety, the first 2 participants in each of the main study cohorts will be dosed (one with REGN17092 and one with placebo) at least 24 hours prior to the remaining participants in the cohort. After these 2 participants complete dosing, the safety data will be collected and reviewed by the study doctor and the sponsor. If both agree that enrolment of the remaining participants in the cohort can start, then the remaining participants in the cohort will receive their doses.

## Expansion Cohort(s)

You may be enrolled into an expansion cohort. For any of the doses of the study drug evaluated in the main study cohorts, an extra cohort that includes more participants may be added for the purpose of obtaining additional data on the safety of the study drug and how much study drug is in your blood to support future studies. The REGN17092 dose(s) administered in the expansion cohort(s) will have been determined to be sufficiently well tolerated to allow further evaluation.

The study doctor or member of the study staff will discuss the procedures and samples needed when you arrive at the clinical study unit. The results of these tests will also be used to check the inclusion and exclusion criteria again and to determine whether you are still eligible to participate in the study.

If you are enrolled into an expansion cohort, you will not need to be admitted to the clinical study unit, but you may be admitted at the discretion of the study doctor. The study doctor may recommend you to be admitted for ease and smooth completion of the study procedures.

## Follow-Up Period

The follow-up period lasts about 12 months (1 year) after the study drug or placebo has been administered. The follow-up period consists of outpatient follow-up visits to the clinical study unit, which are visits for which you do not need to stay overnight and can go home on the same day when all the necessary tests and assessments have been done. You will visit the clinical study unit at least 10 times during this period.

You will be asked about any side effects and medication use since the last visit. If a side effect is still ongoing during the clinical study unit visit, follow-up by the study doctor may be done until resolution or stabilization. If you test positive for the SARS-CoV-2 virus that causes COVID-19 during the follow-up period, you will be asked to inform the study doctor and share your test results as soon as possible.

The study calendar for the study periods, and for each test and procedure that will be performed at each visit, is summarized in tables later in this form. Additional collection times, or changes to or removal of collection times of blood pressure, vital signs, electrocardiogram (ECG), and/or laboratory safety tests, will be permitted as necessary, to ensure appropriate collection of safety data.

# 5. Will I benefit from the study?

As REGN17092 has not yet been administered to humans, there is no evidence that it can provide clinical benefit when administered.

# 6. What are the possible risks and discomforts of taking part?

## 6.1. What are the possible side effects of REGN17092?

Participation in a study involves some risk.

This section provides information about known or possible side effects that may happen when receiving REGN17092. Everyone in the study will be watched for side effects, and you will be

told about any important new safety findings related to the study drug. Talk to the study doctor if you have any questions about the risks described below.

There is currently no information about REGN17092 use in people. However, there is a lot of safety information in people for a drug that is similar to REGN17092. This drug, Ronapreve, also called casirivimab and imdevimab, has been tested to treat and prevent COVID-19. REGN17092 works like this drug and was made in the same way. Since the drugs are similar to one another, the side effects expected from REGN17092 may be similar to what was seen with casirivimab and imdevimab.

#### Risks of receiving REGN17092

For people who receive the drug as an infusion in a vein in the arm, reactions related to the infusion may occur. These reactions may include nausea, chills, dizziness, rash, hives, itchy skin, flushed (red) skin, and fast or shallow breathing. These kinds of reactions were seen in people who received casirivimab and imdevimab.

For people who receive REGN17092 as an injection under the skin, reactions at the injection site may occur. Injection site reactions can include patchy red skin, itchy skin, hives, bruising, fluid build-up, pain, and tenderness. Dizziness or swollen lymph nodes were also seen in people who received casirivimab and imdevimab and may occur with REGN17092.

Allergic reactions may also occur when receiving the drug. It is important to tell the doctor about any prior allergies or allergic reactions. In some cases, severe allergic reactions (anaphylaxis) may occur. Symptoms of a severe reaction can include shortness of breath, sweating, and rapid heartbeat. Severe allergic reactions can be life-threatening. **Get medical help right away** if you think you are having severe symptoms of any kind.

# Other possible risks

Risk of Virus Resistance to Treatment

There are now many variants (types) of the virus that causes COVID-19. REGN17092 is designed to work against variants, including Delta and Omicron. However, there is a risk that the drug could work less well, or could be ineffective, against future variants.

Risk of Unwanted Immune Response

Antibodies are a part of the body's normal defense mechanism against a foreign substance and, as such, the body could make its own antibodies against REGN17092. If this were to occur, this could make the drug work less effectively or cause side effects similar to allergic reactions or side effects that are not known at this time. This has not occurred often in people who received a similar drug (casirivimab and imdevimab).

Possible Risk of the Study Drug Interfering with Vaccines or Fighting Off a Future Infection

It is possible that REGN17092 could interfere with your body's response to COVID-19 vaccines. It could also interfere with your body's ability to fight off a future infection of the virus that causes COVID-19.

VV-RIM-00310795-1.0 Approved - 01 Aug 2023 GMT-5:00

# Possible Risk of Virus Infection Getting Worse

Treatments containing antibodies can sometimes make it easier for a virus to cause infection. If this happens, symptoms could get worse weeks to months after receiving the drug. Participants will be watched for negative outcomes like this. In people who received a similar drug (casirivimab and imdevimab), there has been no evidence of this side effect happening.

Risks Related to Pregnancy and Breastfeeding

Antibodies like REGN17092 may cross the placenta (the lining around a fetus during pregnancy) or get into breast milk. Because of this, it is possible that the drug could travel from a mother to a developing fetus or newborn baby.

It is not known if the drug may harm a pregnant mother or baby during pregnancy or breastfeeding, or whether the pregnancy could be lost. Studies with a similar drug (casirivimab and imdevimab) have included women who were pregnant or became pregnant during the study. In these individuals, no safety concerns have been seen.

If you are pregnant or breastfeeding, or plan to become pregnant during the study, you will not be allowed to participate in the study.

#### Unknown Risks

There may be other side effects related to REGN17092 that are unknown at this time. Some of these unknown side effects could be serious or life-threatening.

It is important that the study doctor or staff are told right away about any side effects or health changes. It is also important to report the use of any new medicine or supplements, including vitamins, herbal remedies, over-the-counter drugs, or prescription drugs.

# 6.2. What are the possible risks or discomforts of the examinations during the study?

The examinations of the study may cause the following discomforts and risks:

#### Testing for Infection by the Virus that Causes COVID-19

As part of the study, you will be tested at screening to see if you have the virus that causes COVID-19. One of the methods below may be used to collect the sample for testing. If a swab method is used, more than one swab may be collected. Before you sign this form, you will be told how the test sample will be collected.

**Nasopharyngeal (NP) Swab:** This method involves taking a sample at the back of your throat. A swab is gently inserted about three inches into the nose until it reaches the throat. The swab is rotated a few times and then removed. This may be done in one or both nostrils.

**Oropharyngeal (OP) Swab:** This method is similar to an NP swab. A sample is taken at the back of the throat, but the swab is inserted through the mouth. The swab is rotated a few times and removed.

**Nasal Swab:** A nasal swab involves taking a sample on the inside of 1 or both of your nostrils. The swab is inserted about 1 inch or less into your nose, rotated a few times, and removed. This may be done in 1 or both nostrils.

**Saliva:** A saliva sample is taken by spitting into a specially designed cup several times until enough saliva is collected.

R17092-HV-2312 Main ICF Version 2.0

The risks of the test are minimal. Samples taken from the back of the throat (NP and OP swabs) are more likely to be uncomfortable. They may cause you to gag or feel the urge to sneeze or cough. An NP swab may give you a minor nosebleed. Nasal swabs and saliva samples have little risk of being uncomfortable.

You will be told if you test positive for the virus that causes COVID-19.

#### Nasal Fluid:

Nasal secretions may be obtained by inserting a nasal sponge into the nostrils for up to 10 minutes. Minor discomfort in the nostrils and nosebleed may happen after this is done.

Nasal fluid may be collected during the treatment and follow-up periods.

# Blood Sampling/Placement of Intravenous Catheter:

Blood will be taken to check your health and carry out the research goals described in this form. Drawing blood from your arm may cause pain, bleeding, bruising, or infection localized around the injection site. Similarly, some participants may feel dizzy or even faint during the procedure. The study staff who takes the blood will do all they can to keep these discomforts to a minimum.

The total amount of blood drawn will vary at each visit. Over the course of the study, about 384 mL of blood will be taken in total (a standard blood donation, for example, the Red Cross, contains 470 mL of blood).

You may need to have visits that are not currently planned as part of the study. These unplanned visits may be needed if you think you have symptoms of COVID-19. These unplanned visits may also be needed to check on side effects, repeat laboratory tests, or for other reasons that will be explained to you before the visit. These visits could include having blood and/or nasal or saliva samples taken. Repeat or unscheduled blood samples will not exceed 50 mL; these amounts involve no risk for your health.

#### Infusion or Injection:

You will be given a single dose of the study drug (REGN17092) or placebo either as an under the skin injection or as an infusion in a vein.

Any time you receive an infusion, you may experience brief pain, bleeding, bruising of the skin, soreness, swelling, and possible infection at the infusion site. Injections under the skin can cause pain, tenderness, redness, itchiness, swelling, or warmth where the injection is given.

In addition to these general risks of infusion and injection, other side effects may happen because of the study drug itself. These risks are described above in Section <u>6.1</u> (What are the possible side effects of REGN17092?).

### Vital Signs:

The study staff will take your vital signs, which may include measuring your blood pressure, pulse rate, breathing rate, and temperature in a lying, seated, or standing position. Taking your blood pressure measurements requires wrapping and then inflating a blood pressure cuff, usually around one of the arms. You may experience mild discomfort in your arm while the cuff is inflated.

# **Urinalysis:**

Your urine will be collected during screening. You will be provided a container to collect your urine sample in and the study staff will collect the container from you.

# **Electrocardiogram**:

You will be asked to have an electrocardiogram (ECG) done at certain points in the study. This test records electrical activity of your heart and is done to evaluate your heart rhythm before, during, and after you are given the study drug or placebo. For ECG recordings, a few sticky patches, called electrodes, will be placed on your chest. The attachment of the patches and removal of these patches from the skin may cause a reversible skin reaction such as redness or itching. You may also experience localized skin discomforts and/or hair loss at the location of the lead placements.

#### Physical Examination:

Your doctor will perform a physical exam to check your overall health several times during the study. This examination will include measuring your weight (at screening and pre-dose on day 1) and height (at screening). A physical examination and having your weight measured may make you feel uncomfortable.

#### **Pregnancy Test:**

If you are a woman who is able to have children, you will have to have blood or urine pregnancy tests during the study.

Blood draws may cause discomfort, bruising, or infection at the site where blood was taken. Some people become faint or dizzy when giving blood. Collecting your own urine may make you feel uncomfortable.

# 6.3. Can I take other medicines during the study?

The use of prescription and non-prescription medication is generally not allowed during this study. Do not hesitate to ask your study doctor for more explanation about the use of other medicines and food supplements.

# 6.4. Will my participation in the study have an <u>impact on my daily activities</u>?

Any strenuous exercise should be avoided during the study. You will not be allowed to donate blood or have planned, elective surgeries during the study.

### 6.5. Can my partner or I get <u>pregnant</u>, or can I breastfeed during the trial?

This section is intended solely for participants with a potential to become pregnant or participants who may get their partners pregnant.

#### Female Participants:

You will not be allowed to take part in this study if

- you are pregnant,
- you wish to become pregnant in the near future, or

R17092-HV-2312 Main ICF Version 2.0

• you are breastfeeding.

Egg/ovum donation is also not allowed during the study and for up to 12 months after the last dose of REGN17092 or placebo. Please discuss this point with the study doctor if this applies to you.

If you take part in the study, and you are a woman of childbearing potential, you must use one of the following authorized methods of contraception, during the study and for 12 months after the last dose of REGN17092 or placebo:

- Stable use of combined (estrogen- and progestogen-containing) hormonal contraception (oral, intravaginal, transdermal) or progestogen-only hormonal contraception (oral, injectable, implantable) started at least 2 or more menstrual cycles prior to screening
- Intrauterine device (IUD) or intrauterine hormone-releasing system (IUS)
- Bilateral tubal occlusion/ligation
- Vasectomized partner (provided that the male vasectomized partner is your sole sexual partner and has obtained medical assessment of surgical success for the procedure)
- And/or sexual abstinence

Please discuss the contraception methods with your study doctor if this applies to you. Please inform the study doctor in case you would decide during the study to change your method of contraception. You will not be reimbursed by the sponsor for any contraception you take during the study.

You will be required to have a pregnancy test during the screening period, at the start of the study before the first dose of REGN17092 or placebo, at 3 visits during the follow-up period, and at the end of the study.

Nevertheless, if you become pregnant during the study, you should inform the study doctor and your treating physician immediately. The study doctor will follow up with you about your pregnancy. Only information regarding your pregnancy will be shared with the sponsor. No identifying information will be given to the sponsor. By signing this consent form, you agree to this follow-up.

# Male Participant:

Taking REGN17092 could have an effect on your sperm and could lead to an unknown risk for an unborn child.

If you take part in the study, you should not donate sperm during the study and for 12 months after the last dose of REGN17092 or placebo. Please discuss this point with the study doctor if this applies to you. If you participate in the study, you must use medically acceptable birth control (male latex condom) for 12 months after receiving the study drug or placebo injection or infusion, unless your partner is unable to become pregnant (for example, if your partner is medically sterile or you have had a vasectomy) or you practice sexual abstinence.

You must commit to inform your female partner of your participation in this study and of the potential risk to an unborn child.

R17092-HV-2312 Main ICF Version 2.0

Nevertheless, if your partner becomes pregnant during the study, you should immediately inform the study doctor. If you agree, (s)he will contact your partner to ask her to be followed up during her pregnancy and its outcome and to sign a specific informed consent (for the pregnant partner).

# 7. What if something goes wrong within the trial?

Even if there is no fault, the sponsor is liable for harm caused to you whether directly or indirectly related to your participation in the study. The sponsor has taken an appropriate insurance (a so-called "NO FAULT INSURANCE") for this liability. A copy of the insurance certificate can be obtained from the study doctor or study staff.

If you (or in the event of death, your rightful claimants) seek compensation for a harm to your health as a direct or indirect result of participating in the study, you must inform your study doctor or study staff promptly.

If the study doctor believes that a link between the new or worsened health problem(s) and the study is possible, he/she will inform the study sponsor. The sponsor will then immediately initiate the declaration procedure to its insurance company. If the company considers it necessary, it will appoint an expert to assess whether there is a link between your reported health problem(s) and the study.

Whenever you feel it is appropriate, or if you or your rightful claimants disagree either with the study doctor or with the expert appointed by the insurance company, you may contact the insurance company, or proceedings may be brought against the insurance company. You will find the contact details on the front page of this form.

# 8. What if other treatment options or new information on REGN17092 become available during the course of the study?

During the course of the study, important new information might become available, possibly affecting your decision to (further) participate. For example, important new information on REGN17092 may become available. It is the duty of the study doctor to discuss this new information with you and to give you the opportunity to reconsider your participation in the study.

# 9. Can my participation in the study end prematurely?

As explained in detail below, your participation in the study may end prematurely when

- you decide to withdraw your consent,
- the study doctor decides to end your study participation, or
- other entities interrupt or end the study.

In any case, if your study participation ends prematurely, the study doctor will discuss your future medical care with you. The sponsor can continue to retain and use any data that have already been collected before the end of your participation. This is to avoid skewing/biasing results of the study (as described in Section 11.4, page 16).

If you experienced a side effect at the moment of stopping REGN17092 or placebo, the study doctor may contact you in the future to see if it has resolved or not after the end of the study participation.

If you experience a new side effect after the end of your study participation, you may contact the study doctor to ask for a follow-up.

#### 9.1. You decide to withdraw your consent

You are entitled to withdraw your consent for any reason, at any time, without having to justify your decision. However, for your safety, you should inform the study doctor of your decision. Although it is not mandatory, it may be useful for the study doctor and for the sponsor to know the reason of your decision (for example side effects, frequency of clinical visits).

If you withdraw your consent, this means you decide to stop

- the treatment with REGN17092 or placebo, and
- all study-related visits and examinations.

Please discuss with your study doctor to evaluate the process of your withdrawal (in light of your situation), including any follow-up visits or procedures.

In any case, no new data will be sent to the sponsor.

If your biological samples (eg, blood samples, urine samples) have already been used or analyzed before the withdrawal of your consent, the Regeneron Parties still have the right to use the results from those tests.

The biological samples that have been collected (but not tested) before the withdrawal of your consent, and the data obtained from it, can also still be used by the Regeneron Parties. You may ask for a destruction of those samples.

### 9.2. The study doctor decides to end your study participation

The study doctor may end your study participation because:

- you become pregnant during the study,
- it is better for your health,
- he/she determines that you are not following the instructions given to participants, or
- any other reason that will be explained.

# 9.3. Other entities may interrupt or end the study

The sponsor and the competent Belgian health authorities may interrupt or end the study because:

- REGN17092 causes more (serious) side effects than anticipated, or
- any other reason that will be duly motivated by such party.

VV-RIM-00310795-1.0 Approved - 01 Aug 2023 GMT-5:00

# 10. Will my participation in the study involve extra costs for me?

#### 10.1. Examinations and treatments paid by the sponsor

The sponsor has arranged to compensate the hospital or clinical study unit for:

- the time devoted to the study by the study doctor and the study staff,
- the visits/consultations and all scheduled examinations specific to the study,
- the investigational treatment (REGN17092 and any other medication and material specifically used for the study).

This study is conducted in healthy volunteers, and therefore all the treatments or examinations you will undergo are study-specific and will be paid for by the sponsor and will not be charged to you.

If you need more details, please contact the study staff.

The visits and treatments which are a consequence of a side effect are also considered as study-specific.

## 10.2. Other expenses paid by the sponsor

If you decide to take part in this study, this will not involve any extra costs for you for the study doctor's time or certain procedures and supplies related to this study. The visits and procedures identified as specific to the study, in the description of the course of the study in Section 4, page 4, will be paid for by the sponsor.

You will receive payment for your participation in the study. You will receive half of the payment after the day 120 visit, and the rest of the payment upon completion of the entire study. Total financial compensation is as follows:

- €2722 Euro if you were enrolled in a main cohort with IV administration (into a vein)
- €2786 Euro if you were enrolled in a main cohort with SC administration (under the skin)
- €2380 Euro if you were enrolled in an expansion cohort with IV administration
- €2358 Euro if you were enrolled in an expansion cohort with SC administration

Compensation may be pro-rated based on the portion of the study completed.

If based on newly available data, you are asked for extra visits during the study, these may be compensated based on the duration of the visit.

Please note that if you withdraw from the clinical study for non-medical reasons or for reasons not confirmed by the study doctor, you may be paid pro-rata. If you are withdrawn from the study for medical reasons related to the study, having received study medication, you will receive payment in full.

If you are a 'back-up' or 'reserve' participant, you will receive a compensation of €484 euros if you are in a main study cohort or €433 euros if you are in an expansion cohort, including transport and parking costs. A back-up participant is a participant who qualifies to participate in

the study and is admitted to the unit as a reserve participant. This means that if another participant is excluded from the trial prior to being dosed, the back-up participant is expected to be able to take the participant's place in the study for the duration of the trial. In this case, you will be expected to participate in all study visits as described and you will be reimbursed for the entire study. However, if you are not asked to take another participant's place, you can leave the unit once all other participants have been dosed and will be reimbursed the renumeration of a back-up participant.

If based on newly available data, you are asked for extra visits during the study, these will be compensated with €70 euros per visit. If based on newly available data the in-patient stay is prolonged, you will be compensated with €255 euros for every additional 24-hours stay.

The study staff will contact you for the practical arrangements.

Your biological samples are deemed to be a "donation". You will not receive any financial benefit associated with the development of new therapies derived from the use of your biological samples, which may end up having commercial value.

# 11. Which data are collected about me during the study and what will happen with them?

## 11.1. Which data are collected and processed during the study?

The collected and processed personal data concern information about your health and medical condition. This includes your medical history, some of your background information (eg, your age, sex, and ethnic origin) and the results of examinations required by the study.

# 11.2. How will the study doctor treat my personal data?

The study doctor is bound by professional secrecy about the data collected.

This means that he/she will never reveal your identity, including in a scientific publication or a lecture, and that he/she will encode your data (*that is* by replacing your identity by an identification code in the study) before sending them to the sponsor.

Therefore, the study doctor and the study staff, under the responsibility of the study doctor, will be the only ones able to establish a link between your identity and the data transmitted during the study, with the exceptions listed under Section 11.6.

The data transmitted to the sponsor will not allow the sponsor to identify you.

#### 11.3. What will happen to information about me collected during the study?

Your participation in the study means that your personal data

- are collected by the study doctor, and
- are used in an encoded form by the Regeneron Parties.

The study doctor and the Regeneron Parties can only use the encoded personal data for research purposes, in connection with scientific publications within the context of the study that you participate in, or for a broader use of the encoded data if described below.

In addition, the sponsor may grant external researchers (not involved in this study) access to the encoded data.

### 11.4. How will my data be handled?

Your study data will be processed in accordance with the General Data Protection Regulation (GDPR) and the Belgian law on data protection of 30 July 2018. The sponsor is responsible for this processing.

Processing your personal data in this study is allowed because we are conducting scientific research, and the sponsor has a legitimate interest to ensure high standards of quality and safety to its medicines.

# 11.5. Do I have access to my data collected and processed during the study and can I rectify them?

You are entitled to ask the study doctor what data are being collected about you and how those data will be used in connection with the study.

You have the right to

- inspect and access these data,
- request that your data be erased,
- ask for correction if they are incorrect,
- restrict the processing of your data,
- object to the processing of your personal data,
- withdraw your consent for the processing of your personal data.

However, these rights may be limited or postponed due to regulatory requirements and to preserve scientific integrity, as the data must be managed in specific ways in order for the research to be reliable and accurate. Note that personal data collected before withdrawal of consent will continue to be used to avoid skewing of results in the study. However, no new information will be collected about you without your consent.

#### 11.6. Who, other than the study doctor and study staff, has access to my personal data?

To verify the quality of the study, it is possible that your personal, uncoded data or information in your medical records relevant for the study will be examined by people outside the study staff, but under the responsibility of the study doctor directly at the study site. These persons must be subject to professional secrecy or a confidentiality agreement. The following might be considered:

- the personnel designated by the sponsor of the study (MONITORS and AUDITORS), and people or organizations providing services for or collaborating with the sponsor. They will however never transfer your name and contact details to the sponsor.
- inspectors of competent health authorities worldwide
- an independent audit group

R17092-HV-2312 Main ICF Version 2.0

• people designated by the Ethics Committee

For the needs of the study, the <u>encoded</u> study data may be sent to other European Union (EU) and non-EU countries and may be reviewed by:

- personnel (other than the inspectors) of competent health authorities of Belgium (Federal agency for medicines and health products, FAMHP) and other EU and non-EU countries,
- the evaluating Belgian Ethics Committee(s),
- external researchers,
- the sponsor of the study, personnel designated by the sponsor, and people or organizations providing services for or collaborating with the sponsor, and/or
- group companies of the sponsor in Belgium, and in other EU and non-EU countries.

Regeneron is based in the United States (US), and your encoded personal data may be accessed from or transferred to locations where Regeneron operates, which includes the US, Canada, United Kingdom (UK), and EU member states. Your encoded personal data may also be transferred to other countries where Regeneron has a collaborator or where it seeks to market its products. Although your encoded personal data may be transferred outside of your country where data protection laws may differ, Regeneron will take measures to ensure your encoded personal data and your rights are adequately protected in accordance with the law.

The European regulation and the Belgian legislation on data protection have requirements for transferring data to non-EU countries. The sponsor must ensure equivalent guarantees regarding personal data protection standards before transferring the encoded data to non-EU countries. If for this purpose, there is a data protection agreement, a copy of this agreement may be obtained via the study doctor. You can always contact your study doctor to obtain more information about any such transfers.

### 11.7. What will happen to the results of the study?

In order to further medical science, your study data and results may be provided to qualified researchers who request it for legitimate research purposes. Data and results from this study will also be presented at meetings or published in journals. While your study data may be shared with these researchers or publications, direct identifiers (such as your name) will not be shared with these researchers and will not be in any presentation or publication. A description of the study and its results may be published in medical journals once the study is over. You may request a copy of the publication, or a summary in plain language, from the study staff. A description of the study will also be available on <a href="https://euclinicaltrials.eu/and/or">https://euclinicaltrials.eu/and/or</a><a hre

number given on the front page of the informed consent form. The websites will include a summary of the results within 1 year after the end of the study.

These websites or publications will not include information that can identify you.

## 11.8. Will my data be used for other purposes than for the study in which I take part?

The results of the study will be used to conduct the research described in this form. As advancements in medical technology continue, Regeneron, its collaborators or those developing the study drug, and their affiliates, representatives, agents, and contractors (the "Regeneron Parties") may reanalyze the study data and the results in future research projects to find new scientific information about the study, study drug, COVID-19, or other related diseases.

Any additional or future research outside of the research described in this consent form must always be approved by a recognized Belgian Ethics Committee.

## 11.9. How long will my data be kept?

After the end of the study, your encoded data will be retained for at least 25 years to conduct and ensure the validity of the research. This will also be the case if you stopped study participation prematurely.

If you withdraw your consent to take part in the study, to guarantee the validity of the research and due to regulatory requirements, the data encoded up to the point at which you withdraw will be retained. No new data may be sent to the sponsor.

# 12. Which biological samples are collected from me during the study and what will happen with them?

# 12.1. Which biological samples are collected from me during the study?

Biological samples are samples of human body material (for example blood, tissue, urine, fecal stool). In this study, the following biological sample(s) may be taken:

- blood
- urine
- saliva
- nasal fluid, and
- nasopharyngeal/oropharyngeal/nasal swabs.

You may not directly benefit from biological sample testing in this study, since it may take several years for results to become available. However, it is possible that the treatment of future patients can be improved based on what we learn from studying biological samples in this study. Please note that if you consent to participate in the study, biological samples will be collected.

#### 12.2. What will happen to the collected biological samples?

The collected biological samples will be managed and stored at Regeneron, Tarrytown, USA, or at a storage facility designated and supervised by Regeneron in the US. Unused samples will be destroyed.

Your blood and nasal fluid samples will be collected and used by Regeneron Parties to support the current study objectives and may be used for research by the Regeneron Parties. This includes submitting study results to public health agencies for study drug approval, when

R17092-HV-2312 Main ICF Version 2.0

applicable. During the study and for up to 15 years after the study closes, your samples will be used for the following goals:

- how the study drug works in the body,
- why some people respond better to the study drug,
- why some people have reactions to the study drug,
- better understanding of COVID-19,
- developing diagnostic tests related to the study drug and COVID-19, and
- understanding the prevention and treatment of COVID-19.

You have the right to take back your consent to having these samples used and stored. If you would like to have your samples destroyed, you can contact the study doctor in writing or verbally notify them. The study doctor and Regeneron Parties will take reasonable steps to destroy them. Please understand that if your samples have already been tested, the results cannot be erased and will be available to the Regeneron Parties even after your samples are destroyed. If you leave the study, but do not take back consent to use and store your samples, the samples will continue to be used as described above.

#### 12.3. How will my biological samples be handled?

The procedure to encode your biological samples is the same as that used for your personal data (see Section 11.3, page 16). Samples sent to the sponsor or to organizations working in collaboration with the sponsor, will only be labelled with your study identification code (i.e., Participant ID).

As part of the study, the sponsor might transfer (a part of) your samples to a laboratory that is working with them. This laboratory may only use your coded samples as specified in this document. Samples will always contain the participant ID to ensure traceability by the sponsor.

Your biological samples are deemed to be a "donation." You will not receive any financial benefit associated with the development of new therapies derived from the use of your biological samples, and which may have commercial value.

# 12.4. What happens with any <u>remainders</u> of biological samples once the analyses described in this document have been carried out?

The sponsor shall use the biological samples within the context of the study as described above.

# 12.5. Will any <u>additional</u> biological samples be collected and used for additional research?

In this study, no additional biological samples outside of the scope of research described above will be collected.

# 13. Who has reviewed and approved the study documents?

The documents of the study have been reviewed by:

- the Belgian competent health authorities (FAMHP) or if applicable by the competent national health authorities of other EU members states and
- an independent Belgian Ethics Committee.

It is the task of the competent health authorities and the Ethics Committees to protect people who take part in a study. The health authorities will ensure that the study is conducted in accordance with the applicable legislation.

You should not, under any circumstances, take their approval as an incentive to take part in the study.

# 14. What happens in case of incidental findings?

If by chance, and in addition to the study objectives, a result is discovered during the study that may be important to your health or the health of your blood relatives (called "incidental findings"), the sponsor may inform the study doctor.

Certain results produced as part of this study are for research purposes only. The results are not reviewed for medical diagnosis of any disease. Because the results obtained during the course of the research have only clinical research value and are not for medical diagnosis, the sponsor generally does not provide individual results to you. In some circumstances, the sponsor may provide certain results to your study doctor. If, during the course of the study, the study doctor learns information related to your health from the study procedures, the study doctor may discuss this information and your options with you. If this occurs, with your consent the study doctor will notify you and your treating physician about your results and potential consequences. If necessary, the study doctor and/or the treating physician will advise you on the next steps.

You agree or disagree to being informed of incidental findings by ticking the appropriate checkbox in Chapter II, page 23.

Information, you can contact the sponsor's Data Protection Officer at <a href="DataProtection@Regeneron.com">DataProtection@Regeneron.com</a>. Please be aware that because the sponsor only maintains coded study data, it generally cannot respond directly to individual requests about your privacy rights. Therefore, you should address any of these requests regarding the following rights to the study site; see contact details on page 2. If you have any questions relating to how your data are being processed, you may contact the study doctor. The data protection officer in your hospital can be contacted as well (see contact details on page 2). If you have any questions regarding your rights as a participant in the study, you can contact the ombudsman service in your hospital on the telephone number: +32 16 34 48 18. If necessary, the ombudsman service can put you in touch with the Ethics Committee.

Finally, if you have a complaint concerning the processing of your data, you can contact the Belgian supervisory authority who ensures that privacy is respected when personal data are processed.

# **REGENERON**

The Belgian supervisory authority is called:

Data Protection Authority (DPA) Drukpersstraat 35, 1000 Brussels Tel. +32 2 274 48 00

e-mail: contact@apd-gba.be

Website: https://www.dataprotectionauthority.be

#### **CHAPTER II - INFORMED CONSENT**

# **Participant**

## PREREQUISITES FOR YOUR PARTICIPATION IN THE STUDY

- I declare that I have been informed of and that I understand the purpose of the clinical study, its duration, possible risks and discomforts, the precautions that I have to take, and what is expected of me. My rights have been explained to me and I have understood those rights.
- I have had enough time to think about taking part in this study and to discuss it with a trusted person (for example friends, relatives, treating physician, etc).
- I have had the opportunity to ask any questions that came to mind and have obtained a satisfactory response to my questions.
- I understand that my participation in this study is voluntary and free from any coercion and that I am free to stop my study participation at any time.
- I understand that data about me will be collected and that they will be treated confidentially.
- I understand that by participating in the study, my personal data will be processed as described in this consent form.
- I understand that the sponsor has taken out an insurance in case I should suffer any damage in connection with my participation in this study.
- I understand that when participating in this study, I will not have any costs.
- I agree to my treating physician(s) being informed of my participation in this study.
- If I participate in another interventional study, I must let the study doctor or study staff know. I agree that I will not participate simultaneously in another interventional study (eg, with a study drug, medical device, experimental surgical techniques) without informing the study doctor or study staff, and that participation in this study or continuation of participation in this study may be refused if justified.
- I understand that I need to cooperate and follow the study doctor's and study staff's instructions regarding the study.
- I understand that participation in the study might end for me without my consent if I need other treatment, do not follow the study plan, have a study-related injury, or for any other justified reason.
- I certify that all the information I have given about my medical history is correct. I understand that my failure to inform the study doctor or designee about any exclusion criteria may harm myself.

# OPTIONAL CONSENTS WHICH ARE NOT A PREREQUISITE FOR YOUR PARTICIPATION IN THIS STUDY.

| 1. | 1. As described in Chapter I, Section 14, page 20, it may happen that incidental findings a discovered by the study doctor that may be important to your health or the health of yo blood relatives. | |
|---|---|---|
| | If this happens: do you want the study doctor physician) of this result? | to inform you (directly or via your treating |
| | (Tick as appropriate. If you leave this ques want to be informed'.) | tion open, we assume the answer is 'yes, I |
| | ☐ No, I do not want to be informed | ☐ Yes, I want to be informed |

I consent to take part in the study, with the above restrictions, and I have received a signed and dated copy of all pages of this document.

Participant's surname and first name:

Date (DD/MMM/YYYY):

Participant's signature:

# **Investigator (study doctor)**

I, the undersigned investigator, confirm that:

- the participant has been verbally provided with the necessary information about the study, has been explained the content, and has been given an original signed document.
- I have verified that the participant has understood the study.
- I have given the participant sufficient time to agree to take part and to ask any questions.
- no pressure was applied to persuade the participant to agree to take part in the study.
- I operate in accordance with the ethical principles set out in the latest version of the "Helsinki Declaration," the "Good Clinical Practices," and the Belgian Law.

| Investigator's delegate, surname and first name: □ Not Applicable |
|--------------------------------------------------------------------|
| Investigator's delegate, qualification: |
| Date (DD/MMM/YYYY): |
| Investigator's delegate signature: |
| Investigator's, Surname and first name: |
| Date (DD/MMM/YYYY): |
| Investigator's signature: |

A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of REGN17092, an Anti-SARS-CoV-2 (COVID-19) Monoclonal Antibody, in Adult Healthy Volunteers

# **CHAPTER III- STUDY CALENDARS**

Additional collection times, or changes to or removal of collection times, of blood pressure, heart and respiratory rate, electrocardiogram (ECG), and/or laboratory safety tests will be permitted, as necessary, to ensure appropriate collection of safety data.

# STUDY CALENDAR: SCREENING PERIOD (BEFORE YOU START ANY TREATMENT)

| Test or Procedure | During the 28 days before<br>you are first given<br>REGN17092 or placebo |
|---|---|
| Estimated duration of study visit in hours | 1-3 |
| The study doctor will ask for your consent to join the main study, and will check to see if you are eligible for the study | X |
| The doctor will collect some personal information and your medical history | X |
| The doctor will ask about medications you are currently taking and/or any procedures you have had | X |
| The doctor will ask questions about any current symptoms you might be having | X |
| You will be tested for hepatitis B virus (HBV), hepatitis C virus (HCV) and Human Immunodeficiency virus (HIV) | X |
| A physical examination will be done | X |
| Your height and weight will be measured | X |
| Your temperature, respiratory rate, heart rate, and blood pressure will be measured | X |
| An electrocardiogram (ECG) will measure your heart's activity | X |
| Blood will be taken to check your health and check for pregnancy (if you are a woman and able to have children) or to check for a hormone which controls the menstrual cycle in women who are not able to have children | X |
| A urine sample will be taken to check your health | X |

| The doctor will verify if you are negative for the SARS-CoV-2 virus or take an appropriate sample to confirm whether or not | Y |
|---|---|
| you have SARS-CoV-2 virus <sup>1</sup> | 21 |

<sup>&</sup>lt;sup>1</sup> An appropriate sample can be a nasopharyngeal, nasal, oropharyngeal swab or saliva.

# STUDY CALENDAR: TREATMENT

| Test or Procedure | | | | |
|---|---|---|---|---|
| Study Day | | 2 | | |
| | Pre-Dose | Dose | Post-Dose | |
| The study doctor will check to see if you are still eligible for the study | X | | | |
| You will be admitted into the clinical study unit <sup>1</sup> | X | | | |
| The doctor will ask about medications you are currently taking and/or any procedures you have had | X | | | |
| Your weight will be measured | X | | | |
| Your temperature, respiratory rate, heart rate, and blood pressure will be measured <sup>2</sup> | X | | X | X* |
| A physical examination will be done | X | | X | X* |
| The doctor will review any side effects that you have experienced and ask about medications you are currently taking | X | X | X | X* |
| An electrocardiogram (ECG) will measure your heart's activity | X | | X | |
| Blood will be taken to check your health | X | | | |
| A urine sample will be taken to check for pregnancy (if you are a woman and able to have children) | X | | | |
| Blood will be taken to measure the concentration of study drug and run tests to better understand the study drug and how it works <sup>3</sup> | X | | X | |
| Nasal fluid sample may be collected* | X | | X <sup>5</sup> | |
| You will be randomly allocated to receive either REGN17092 or placebo | X | | | |
| Treatment: You will be given a single dose of either REGN17092 or placebo subcutaneously (SC) or intravenously (IV) | | X | | |
| You will be discharged from the clinical study unit <sup>1,4</sup> | | | | X |

<sup>\*</sup>Test or procedure or timepoint not being done in the expansion cohort.

R17092-HV-2312 Main ICF\_Version 2.0

REGENERON CONFIDENTIAL page 28 of 31

<sup>&</sup>lt;sup>1</sup> You will be admitted into the clinical study unit the day before or on the day of dosing at the discretion of the study doctor if you are enrolled in one of the main study cohorts. You will not be required to be admitted to the clinical study unit if you are enrolled into the expansion cohorts, but you may be admitted at the discretion of the study doctor.

<sup>&</sup>lt;sup>2</sup> Your temperature, respiratory rate, heart rate, and blood pressure will be measured at various time points before and after administration of the study drug or placebo.

<sup>&</sup>lt;sup>3</sup> Blood samples will be collected at various time points before and after study drug or placebo administration. The study doctor will inform you when the samples will be collected.

<sup>&</sup>lt;sup>4</sup> If you meet all discharge criteria, you will be discharged from the clinical study unit on day 2, otherwise you will be asked to remain in the clinical study unit based on the study doctor's discretion.

<sup>&</sup>lt;sup>5</sup> Depending on cohort, this collection may be up to 14 hours post-dose.

# STUDY CALENDAR: FOLLOW-UP (AFTER YOUR TREATMENT IS COMPLETED) AND END OF STUDY OR EARLY TERMINATION VISIT

| Test or Procedure | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Study Day | 3 | 8 | 15 <sup>1</sup> | 291 | 45 <sup>1</sup> | 60 <sup>1</sup> | 90¹ | 120 <sup>1</sup> | 2401 | 3651,2 |
| Estimated duration of study visits in hours | 1-2 | 1-2 | 1-2 | 1-2 | 1-2 | 1-2 | 1-2 | 1-2 | 1-2 | 1-2 |
| Your blood pressure and heart rate will be measured | | X | | X | | | | | | X |
| Your temperature and respiratory rate will be measured | | | | | | | | | | X |
| A physical examination will be done | | | | | | | | | | X |
| The doctor will review any side effects that you have experienced and ask about medications you are currently taking | X | X | X | X | X | X | X | X | X | X |
| An electrocardiogram (ECG) will measure your heart's activity | | | | | | | | | | X |
| Blood will be taken to check your health | | X | | X | | | | | | X |
| Nasal fluid sample may be collected* | X <sup>4</sup> | X | | X | | | | | | |
| A serum or urine sample will be taken to check for pregnancy (if you are a woman and able to have children) | | | | X | | | | X | X | X |
| Blood will be taken to measure the concentration of study drug and to run tests to better understand the study drugs and how they work <sup>3</sup> | X | X | X | X | X | X | X | X | X | X |

<sup>\*</sup>Test or procedure not being done in the expansion cohort.

<sup>&</sup>lt;sup>1</sup>Study days are not exact and there is flexibility for rescheduling the visit.

<sup>&</sup>lt;sup>2</sup>You will have an early termination visit if you withdraw your consent or you are withdrawn from the study before the end of the study visit.

<sup>&</sup>lt;sup>3</sup> Depending on the cohort you will be assigned to; the study doctor will inform you when the blood samples will be collected.

<sup>&</sup>lt;sup>4</sup> Day 3 nasal fluid collection for SC cohorts only. Must be performed at least 24 hours after the day 1 post-dose nasal fluid collection.

# **REFERENCES**

- <sup>1</sup> The definition of interventional trial can be found in the Questions and Answers (draft) document of the European Commission which can be found in Eudralex Volume 10, Chapter V which is accessible via the following link: https://ec.europa.eu/health/documents/eudralex/vol-10 en#fragment1.
- <sup>2</sup> This is in accordance with Article 29 of the Belgian Law of 7 May 2004 related to experiments on humans.
- <sup>3</sup> General Data Protection Regulation No 2016/679 of the European Parliament and of the council of 27 April 2016 on the protection of natural persons with regard to the processing of personal data and on the free movement of such data, and repealing Directive 95/46/EC.
- <sup>4</sup> The Belgian Law of 30 July 2018 on the protection of natural persons with regard to the processing of personal data.
- <sup>5</sup> Belgian Law of 19 December 2008 on the acquisition and use of human body material with a view to medical application to humans or scientific research, and the applicable royal decrees.
- <sup>6</sup> In accordance with section 4.3. of the Commission Guideline: Guidance on posting and publication of result-related information on clinical trials in relation to the implementation of Article 57(2) of Regulation (EC) No 726/2004 and Article 41(2) of Regulation (EC) No 1901/2006 (2012/C 302/03). [From the moment the Clinical trial regulation enters into force: In accordance with article 37 of the Clinical trial regulation No 536/2014 of the European Parliament and of the council of 16 April 2014 on clinical trials on medicinal products for human use, and repealing Directive 2001/20/EC; sponsor have to provide summary results of clinical trials in a format understandable to laypersons.]
- <sup>7</sup> In accordance with article 58 of the Clinical trial regulation No 536/2014 of the European Parliament and of the council of 16 April 2014 on clinical trials on medicinal products for human use, and repealing Directive 2001/20/EC.
- <sup>8</sup> Belgian Law of 19 December 2008 on the acquisition and use of human body material with a view to medical application to humans or scientific research, and the applicable royal decrees.
- <sup>9</sup> This is in accordance with Article 21 of the Belgian Law of 19 December 2008 on the acquisition and use of human body material with a view to medical application to humans or scientific research, and the applicable royal decrees.
- <sup>10</sup> When a person of full age is incapable of expressing his will, legal representation must be used which is determined in successive order (administrator, or failing that, the spouse, the legal cohabiting partner, de facto cohabiting partner, an adult child, a parent, an adult brother or sister). The regulation is laid down in article 8 of the law of 7 May 2004 on experiments on the human person.
- <sup>11</sup> Use of an impartial witness is necessary when either the participant or the participant's legally authorized representative speaks and/or fully understands the language of the approved informed consent form but cannot read and write due to any physical impairment or is visually impaired. An interpreter is necessary when the investigator doesn't speak the language of the participant.
- <sup>12</sup> Belgian Law of 7 May 2004 related to experiments on humans, and the applicable royal decrees.